CLINICAL TRIAL: NCT03666065
Title: Diluted Insulin in Young Children: Bigger Volumes for Smaller Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2000023577; 5-ECR-2014-112-A-N (Other Grant/Funding Number: Juvenile Diabetes Research Foundation)
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aspart-U100 Insulin (Active Comparator): Standard Concentration Rapid Acting Insulin
  Interventions: Drug: Aspart insulin
- Aspart-U25 Insulin (Experimental): Diluted Concentration of Rapid Acting Insulin
  Interventions: Drug: Aspart insulin

INTERVENTIONS:
Drug: Aspart insulin — Standard insulin
  Other Names: Standard Concentration insulin

SUMMARY:
The aim of this study is to compare the pharmacokinetic (PK) profile of diluted insulin aspart (U25) with undiluted insulin aspart (U100) in school-aged children and adolescents with type 1 diabetes (T1D) utilizing the euglycemic clamp technique and a standardized meal in a controlled research environment.

The investigators hypothesize that dilution of insulin aspart (U25) will alter the PK properties as compared to undiluted aspart.

DETAILED DESCRIPTION:
Study Design: participants age 9-15 y/o will be enrolled in a randomized cross-over trial, in which each participant will undergo two 24-hour admissions. Each admission will include a meal-study on the evening of admission followed by a euglycemic clamp study performed the following morning. During one of the admissions, participants will use undiluted insulin aspart (U100) while on the other the participants will receive diluted insulin aspart (U25).

(Figure 1)

Participants. 12 participants will be recruited between the ages of 9-15 years, who have had diabetes for at least 6 months' duration, on continuous subcutaneous insulin therapy for at least 1 month and have an HbA1c ≤ 10%. Those with a history of diabetes ketoacidosis (DKA) or severe hypoglycemia in the month prior to enrollment and those with other conditions/medications affecting insulin sensitivity (e.g. metformin) will be excluded from the study.

Study drugs: Diluted insulin U25 will be formulated by adding diluent, which will be obtained from Novo Nordisk, with insulin aspart. The diluted insulin will be formulated by the investigational pharmacy.

Study procedures:

1. Enrollment Visit: The study will be explained to potential participants who meet eligibility criteria and informed consent will be obtained. Demographic data will be recorded and history and physical exam will be performed. HbA1c, hematocrit and urine pregnancy tests in female participants who could become pregnant will be measured to confirm eligibility. Participants will be randomized for the first admission to either diluted insulin studies followed by a second admission for undiluted insulin studies or vice versa.
2. 1st Inpatient Standard Meal Study and Euglycemic Clamp Study: Participants will be admitted to the research unit in the afternoon on the day before the clamp procedure. The participants will be asked to change their infusion set and use the insulin provided for the study procedures- either the diluted or standard concentration insulin, based on randomization at enrollment. On the admission with diluted insulin, pump settings will be adjusted to account for the dilution (increased by a factor of 4 for basal rates, correction factors, and carbohydrate ratios). An intravenous catheter will be inserted into antecubital vein for blood sampling. Once the IV is placed, Yellow Springs Instrument (YSI) glucose values and insulin levels will be obtained at least every half hour.

   At dinner (~6p.m.), participants will receive a meal prepared in the metabolic kitchen to allow for accurate determination of carbohydrate, fat and protein content. Participants will be asked to estimate the carbohydrate content of the meal prepared by the metabolic kitchen. The participant will bolus just prior to the start of the meal based on the carbohydrates estimated and the pre-meal glucose levels.

   Glucose will be measured by YSI and aspart levels will be measured using the Mercodia iso-insulin enzyme-linked immunosorbent assay. Samples will be taken before the meal and every 10 minutes after the start of the meal for the first hour, every 15 minutes for the second hour, and then every 30 minutes for up to 4 hours after the bolus; namely, at 0, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210, and 240 minutes.

   Participants will then have YSI glucose levels obtained at least every hour overnight with titration of insulin doses as needed to achieve targeted control (goal 80-140mg/dL) by 8a.m. A second IV line will be placed for glucose infusion. Once IV access is established and glucose is in the target range, the euglycemic clamp study will be initiated.

   Prior to the start of the clamp, -15 and 0 minute samples will be obtained for baseline plasma glucose and insulin levels.

   At time zero, a bolus of 0.1 U/kg will be administered via the pump. After administration of the bolus, the insulin pump will be disconnected. Plasma aspart insulin will be measured every 10 minutes for the first 120 minutes and then every 15 minutes for up to 240 minutes using the Mercodia iso-insulin enzyme-linked immunosorbent assay. Plasma glucose will be measured at least every 5 minutes for the duration of the clamp study, which will allow for titration of the glucose infusion rate to maintain euglycemia (target 90 +/- 10mg/dL).

   Following completion of the clamp, the participant will be offered a meal and discharged home with standard concentration insulin and their usual pump settings.
3. 2nd Inpatient Standard Meal Study and Euglycemic Clamp Study: Participants will return for a second admission after a minimum of 7 days since the first study.

The participant will receive whichever concentration of insulin not received during their first admission (ie. If first admission is diluted, then second admission will be standard concentration and vice versa).

The remainder of the study procedures are as indicated above. Following completion of the second clamp study, participants will have completed all study related procedures.

ELIGIBILITY:
Inclusion Criteria:

* T1D of at least 6 months' duration
* Aged 9-15 years
* Continuous subcutaneous insulin therapy for at least 1 month;
* HbA1c ≤ 10%
* Normal hematocrit
* Able to give consent

Exclusion Criteria:

* Admission for DKA during the past 4 weeks
* Severe hypoglycemia during the past 4 weeks
* Other conditions/medications affecting insulin sensitivity (e.g. metformin)

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
maximum insulin concentration | 240 minutes
  maximum insulin concentration

SECONDARY OUTCOMES:
Time to peak insulin concentration | 240 minutes
  Time to peak insulin concentration
Mean Glucose Infusion Rate (GIR) | 240 minutes
  Mean Glucose Infusion Rate
GIR Max | 240 minutes
  Glucose Infusion Rate Maximum
Time to GIR Max | 240 minutes
  Time to Glucose Infusion Rate Maximum

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sherr, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No